CLINICAL TRIAL: NCT01834937
Title: A Post Approval Registry: ExAblate Treatment of Metastatic Bone Tumors for the Palliation of Pain
Brief Title: ExAblate Treatment of Metastatic Bone Tumors for the Palliation of Pain
Acronym: BM019-Registry
Status: Terminated | Type: Observational
Why Stopped: Enrollment Difficulties
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Other Study IDs: BM019-Registry; BM019-Registry (Registry Identifier: BM019-Registry)
Record Dates: First submitted 2013-04-12; First posted 2013-04-18 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Pain Resulting From Bone Metastases
Keywords: ExAblate; MRgFUS; Bone Metastases; Pain Palliation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ExAblate MRgFUS (Magnetic Resonance guided Focused Ultrasound Surgery) — Focused Ultrasound Surgery - FUS delivered by ExAblate for the palliation of pain due to bone metastases.

SUMMARY:
The purpose of this enhanced surveillance study ("ESS") is to collect information regarding chronic adverse events that are possibly related to the ExAblate® System ("ExAblate") that are received by InSightec ("InSightec") following PMA approval. This study will examine adverse events reported in patients undergoing the device procedure for the first two years of commercial experience. Other relevant data may be collected as well.

DETAILED DESCRIPTION:
This proposed Registry will be performed in full compliance with all HIPAA rules and their implementations at potential participating sites. All patients planned to undergo the ExAblate procedure in a commercial setting after PMA approval will be offered a consent so they can be included in the ESS. Non-consenting patients will not be included in the ESS. However, information regarding the total number of subjects treated at each participating site with the device will also be collected.

InSightec will set up a (password protected) EDC database for the sites to enter the information of participating subjects treated with the ExAblate device from all U.S. sites using the ExAblate procedure for the bone metastases indication. This will occur for a total duration of 2 years following device approval. It should be noted that any adverse event that meets the Medical Device Report ("MDR") definition will be reported as an MDR as well.

There will be no control group. Reporting to FDA will occur at six-month intervals for the first two-years after PMA approval.

ELIGIBILITY:
This study collects safety data on patient treatments performed commercially under the FDA approved labeling.

* Eligibility is as per approved device indication.
* All registry-consented patients who undergo commercial ExAblate procedure for bone mets palliation after device approval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consented patients from all participating US sites who receive the commercial ExAblate procedure during the first year after approval will be included. This study/registry will examine treatment background information such adverse events, primary cancer type, treatment frequency, etc., reported in patients undergoing the device procedure for the first two years of commercial experience.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Two Years
  This study is designed to collect safety data during the first two years of commercial use of ExAblate MRgFUS treatment for palliation of pain resulting from bone metastases.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - City of Hope, Duarte, California
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Mayo Clinic, Rochester, Minnesota
  - Weill Cornell Medical Center, New York, New York
  - University of Virginia, Charlottesville, Virginia